CLINICAL TRIAL: NCT00005278
Title: Retrovirus Epidemiology Donor Study I (REDS I)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1501
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2008-01

CONDITIONS: Acquired Immunodeficiency Syndrome; Blood Donors; Blood Transfusion; HIV Infections; HIV-1; HIV-2; HTLV-I; HTLV-II; Retroviridae Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Retroviridae Infections

SUMMARY:
To conduct a multicenter epidemiologic study of the human retroviruses HIV-1, HIV-2, HTLV-I, and HTLV-II in volunteer blood donors from areas of the United States that were reportedly at high and medium or low risk for HIV. Also, to determine the prevalence of retrovirus seropositivity in first time blood donors; and the rate of retrovirus seroconversion in repeat blood donors as a measure of incidence of infection; to ascertain risk factors for antibody-positive donors; to characterize the blood donor population by geographic location, age, sex, race/ethnicity, and donation history to permit analysis on prevalence, incidence, and risk factors; to identify recipients of retrovirus-positive blood units and conduct clinical and laboratory follow-up of these recipients; and to establish a blood specimen repository for long-term storage of specimens from study donors and recipients for future testing.

DETAILED DESCRIPTION:
BACKGROUND:

HIV is known to be transmissible by blood, blood components, or plasma derivatives. The risk of contracting HIV infection from blood transfusion has been greatly reduced in the United States by implementing stringent criteria for donor acceptance, HIV antibody screening, and new methods of virus inactivation in coagulation factor concentrates. There are additional human retroviruses, however, that may pose a threat to the safety of the nation's blood supply.

The human T-cell lymphotropic retroviruses share many properties, including a preferred tropism for certain lymphocytes and similar modes of transmission. They also differ significantly from each other and on this basis are divided into two distinct groups: the human T-cell lymphocytropic viruses (HTLVs) and the human immunodeficiency viruses (HIVs). HTLV-I, a transforming virus, is the prototype of the first group (HTLVs). It is associated with adult T-cell leukemia (ATL) and is thought to be involved in a central nervous system disorder referred to as tropical spastic paraparesis. This group also includes HTLV-II, which is associated with a T-cell malignancy different from ATL. A newly isolated human retrovirus, termed HTLV-V, may be the etiologic agent of cutaneous T-cell lymphoma/leukemia, and may also be added to this group. HIV, previously known as HTLV-III or lymphadenopathy virus (LAV), a nontransforming virus, causes acquired immunodeficiency syndrome (AIDS) and is the prototype of the second group (HIVs). New members of this group of nontransforming human retroviruses were isolated from individuals in different countries of Africa. LAV-2, also referred to as HIV-2, was isolated from two AIDS patients in Africa, and the first case of AIDS in the United States caused by HIV-2 was reported in January, 1988. A third member of this group, HIV-3, was detected in Africa.

Although the HTLV family of retroviruses is distinct from the HIV family, both groups of viruses infect human T4 (CD4) lymphocytes preferentially and alter the host's T-cell functions. Whereas HTLV-I or HTLV-II primarily induce transformation and proliferation of T Lymphocytes and cause T-cell lymphoma/leukemia in humans, HIV and HIV-2 induce T-cell cytopathology that leads to depletion of CD4 cells.

The spread of HIV by blood transfusion represents a highly efficient mode of transmission. Blood components from donors with antibody to HIV have been shown to transmit the virus with frequencies of greater than 90 percent. Packed red blood cells, platelets, or fresh frozen plasma are all equally effective in transmitting the virus to recipients. It is highly likely, therefore, that recipients who receive blood from donors with antibody to HIV will themselves become infected with the virus. Fortunately, the likelihood of such an occurrence in the United States is now rare due to the implementation of screening procedures and other safeguards. When the study was initiated in 1989, there was a growing concern, however, that human retroviruses other than HIV might threaten the safety of the United States blood supply.

DESIGN NARRATIVE:

Blood donors were asked to participate in this multicenter study. Seropositive donors were notified of test results, counseled, and invited to join the follow-up study. Data collected during the first interview included such items as possible exposures to persons with retroviral infection, sexual preferences and contacts, marital history, intravenous drug use, occupation, travel, knowledge of AIDS and routes of HIV transmission. At subsequent visits a blood specimen was collected for laboratory testing and an assessment made of changes in behavior to reduce the risk of virus transmission.

To calculate incidence and prevalence rates, each center identified the appropriate study population for analysis purposes in collaboration with the coordinating center. For prevalence calculations, the study population consisted of donors at all centers who indicated that they had never donated blood previously. To calculate incidence, the study population consisted of donors who had donated previously in the same center. The incidence of retroviral infections was assessed annually in years three through five. Clinical follow-up of all subjects concluded 48 months after the beginning of enrollment. A blood profile for each center was required to calculate denominator values for incidence and prevalence determinations. The blood profile, or donor demographic characterization consisted of information regarding total donor volume with respect to donation status; new or repeat donor, and if repeat, the time of last donation; age; sex; and race.

An adjunct to the study was the development of repositories of plasma and cell samples from infected donors and negative controls collected at the same time. A potential byproduct of these repositories will be the ability in future years to retrospectively search the REDS frozen repository file for new retroviruses which may appear in the United States population.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Garratty — American Red Cross Blood Services; Martha Higgens — American Red Cross Blood Services; Edward Murphy — University of California at San Francisco; Catharie Nass — American Red Cross Blood Services; George Schreiber — Westat, Inc.; James Smith — Oklahoma Blood Institute

REFERENCES:
- [Background] Busch MP, Glynn SA, Schreiber GB. Potential increased risk of virus transmission due to exclusion of older donors because of concern over Creutzfeldt-Jakob disease. The National Heart, Lung, and Blood Institute Retrovirus Epidemiology Donor Study. Transfusion. 1997 Oct;37(10):996-1002. doi: 10.1046/j.1537-2995.1997.371098016436.x. PMID 9354816
- [Background] Busch MP, Kleinman SH, Williams AE, Smith JW, Ownby HE, Laycock ME, Lee LL, Pau CP, Schreiber GB. Frequency of human immunodeficiency virus (HIV) infection among contemporary anti-HIV-1 and anti-HIV-1/2 supplemental test-indeterminate blood donors. The Retrovirus Epidemiology Donor Study. Transfusion. 1996 Jan;36(1):37-44. doi: 10.1046/j.1537-2995.1996.36196190513.x. PMID 8607151
- [Background] Zuck TF, Thomson RA, Schreiber GB, Gilcher RO, Kleinman SH, Murphy EL, Ownby HE, Williams AE, Busch MP, Smith JW, et al. The Retrovirus Epidemiology Donor Study (REDS): rationale and methods. Transfusion. 1995 Nov-Dec;35(11):944-51. doi: 10.1046/j.1537-2995.1995.351196110900.x. No abstract available. PMID 8604493
- [Background] Busch MP, Korelitz JJ, Kleinman SH, Lee SR, AuBuchon JP, Schreiber GB. Declining value of alanine aminotransferase in screening of blood donors to prevent posttransfusion hepatitis B and C virus infection. The Retrovirus Epidemiology Donor Study. Transfusion. 1995 Nov-Dec;35(11):903-10. doi: 10.1046/j.1537-2995.1995.351196110893.x. PMID 8604486
- [Background] Korelitz JJ, Busch MP, Williams AE. Antigen testing for human immunodeficiency virus (HIV) and the magnet effect: will the benefit of a new HIV test be offset by the numbers of higher risk, test-seeking donors attracted to blood centers? Retrovirus Epidemiology Donor Study. Transfusion. 1996 Mar;36(3):203-8. doi: 10.1046/j.1537-2995.1996.36396182135.x. PMID 8604502
- [Background] Heneine W, Switzer WM, Busch M, Khabbaz RF, Kaplan JE. Molecular subtyping of human T-cell lymphotropic virus type 2 by single-strand conformation polymorphism analysis. Retrovirus Epidemiology Donor Study Group. J Clin Microbiol. 1995 Dec;33(12):3260-3. doi: 10.1128/jcm.33.12.3260-3263.1995. PMID 8586713
- [Background] Johnson D, Hirschkorn D, Busch MP. Evaluation of four alternative methodologies for determination of absolute CD4+ lymphocyte counts. The National Heart, Lung, and Blood Institute Retrovirus Epidemiology Donor Study. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Dec 15;10(5):522-30. PMID 8548331
- [Background] Korelitz JJ, Williams AE, Busch MP, Zuck TF, Ownby HE, Matijas LJ, Wright DJ. Demographic characteristics and prevalence of serologic markers among donors who use the confidential unit exclusion process: the Retrovirus Epidemiology Donor Study. Transfusion. 1994 Oct;34(10):870-6. doi: 10.1046/j.1537-2995.1994.341095026972.x. PMID 7940658
- [Background] Kleinman SH, Kaplan JE, Khabbaz RF, Calabro MA, Thomson R, Busch M. Evaluation of a p21e-spiked western blot (immunoblot) in confirming human T-cell lymphotropic virus type I or II infection in volunteer blood donors. The Retrovirus Epidemiology Donor Study Group. J Clin Microbiol. 1994 Mar;32(3):603-7. doi: 10.1128/jcm.32.3.603-607.1994. PMID 8195365
- [Background] Busch MP, Laycock M, Kleinman SH, Wages JW Jr, Calabro M, Kaplan JE, Khabbaz RF, Hollingsworth CG. Accuracy of supplementary serologic testing for human T-lymphotropic virus types I and II in US blood donors. Retrovirus Epidemiology Donor Study. Blood. 1994 Feb 15;83(4):1143-8. PMID 8111054
- [Background] Schreiber GB, Busch MP, Kleinman SH, Korelitz JJ. The risk of transfusion-transmitted viral infections. The Retrovirus Epidemiology Donor Study. N Engl J Med. 1996 Jun 27;334(26):1685-90. doi: 10.1056/NEJM199606273342601. PMID 8637512
- [Background] Korelitz JJ, Busch MP, Kleinman SH, Williams AE, Gilcher RO, Ownby HE, Schreiber GB. A method for estimating hepatitis B virus incidence rates in volunteer blood donors. National Heart, Lung, and Blood Institute Retrovirus Epidemiology Donor Study. Transfusion. 1997 Jun;37(6):634-40. doi: 10.1046/j.1537-2995.1997.37697335159.x. PMID 9191825
- [Background] Schreiber GB, Murphy EL, Horton JA, Wright DJ, Garfein R, Chien HC, Nass CC. Risk factors for human T-cell lymphotropic virus types I and II (HTLV-I and -II) in blood donors: the Retrovirus Epidemiology Donor Study. NHLBI Retrovirus Epidemiology Donor Study. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Mar 1;14(3):263-71. doi: 10.1097/00042560-199703010-00011. PMID 9117460
- [Background] Williams AE, Thomson RA, Schreiber GB, Watanabe K, Bethel J, Lo A, Kleinman SH, Hollingsworth CG, Nemo GJ. Estimates of infectious disease risk factors in US blood donors. Retrovirus Epidemiology Donor Study. JAMA. 1997 Mar 26;277(12):967-72. PMID 9091668
- [Background] Ownby HE, Korelitz JJ, Busch MP, Williams AE, Kleinman SH, Gilcher RO, Nourjah P. Loss of volunteer blood donors because of unconfirmed enzyme immunoassay screening results. Retrovirus Epidemiology Donor Study. Transfusion. 1997 Feb;37(2):199-205. doi: 10.1046/j.1537-2995.1997.37297203524.x. PMID 9051096
- [Background] Kaplan JE, Khabbaz RF, Murphy EL, Hermansen S, Roberts C, Lal R, Heneine W, Wright D, Matijas L, Thomson R, Rudolph D, Switzer WM, Kleinman S, Busch M, Schreiber GB. Male-to-female transmission of human T-cell lymphotropic virus types I and II: association with viral load. The Retrovirus Epidemiology Donor Study Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Jun 1;12(2):193-201. doi: 10.1097/00042560-199606010-00014. PMID 8680892
- [Background] Murphy EL, Fridey J, Smith JW, Engstrom J, Sacher RA, Miller K, Gibble J, Stevens J, Thomson R, Hansma D, Kaplan J, Khabbaz R, Nemo G. HTLV-associated myelopathy in a cohort of HTLV-I and HTLV-II-infected blood donors. The REDS investigators. Neurology. 1997 Feb;48(2):315-20. doi: 10.1212/wnl.48.2.315. PMID 9040713
- [Background] Busch MP. [Residual risks of viral transmission by transfusions and projected yields of additional screening tests. Retrovirus Epidemiology Donors Study (REDS)]. Transfus Clin Biol. 1996;3(1):7-11. doi: 10.1016/s1246-7820(96)80007-3. French. PMID 8640316
- [Background] Murphy EL, Glynn SA, Fridey J, Smith JW, Sacher RA, Nass CC, Ownby HE, Wright DJ, Nemo GJ. Increased incidence of infectious diseases during prospective follow-up of human T-lymphotropic virus type II- and I-infected blood donors. Retrovirus Epidemiology Donor Study. Arch Intern Med. 1999 Jul 12;159(13):1485-91. doi: 10.1001/archinte.159.13.1485. PMID 10399901
- [Background] Glynn SA, Schreiber GB, Busch MP, Kleinman SH, Williams AE, Nass CC, Ownby HE, Smith JW. Demographic characteristics, unreported risk behaviors, and the prevalence and incidence of viral infections: a comparison of apheresis and whole-blood donors. The Retrovirus Epidemiology Donor Study. Transfusion. 1998 Apr;38(4):350-8. doi: 10.1046/j.1537-2995.1998.38498257373.x. PMID 9595017
- [Background] Murphy EL, Glynn SA, Fridey J, Sacher RA, Smith JW, Wright DJ, Newman B, Gibble JW, Ameti DI, Nass CC, Schreiber GB, Nemo GJ. Increased prevalence of infectious diseases and other adverse outcomes in human T lymphotropic virus types I- and II-infected blood donors. Retrovirus Epidemiology Donor Study (REDS) Study Group. J Infect Dis. 1997 Dec;176(6):1468-75. doi: 10.1086/514143. PMID 9395356
- [Background] Murphy EL, Bryzman SM, Glynn SA, Ameti DI, Thomson RA, Williams AE, Nass CC, Ownby HE, Schreiber GB, Kong F, Neal KR, Nemo GJ. Risk factors for hepatitis C virus infection in United States blood donors. NHLBI Retrovirus Epidemiology Donor Study (REDS). Hepatology. 2000 Mar;31(3):756-62. doi: 10.1002/hep.510310329. PMID 10706569
- [Background] Ownby HE, Kong F, Watanabe K, Tu Y, Nass CC. Analysis of donor return behavior. Retrovirus Epidemiology Donor Study. Transfusion. 1999 Oct;39(10):1128-35. doi: 10.1046/j.1537-2995.1999.39101128.x. PMID 10532608
- [Background] Glynn SA, Kleinman SH, Schreiber GB, Busch MP, Wright DJ, Smith JW, Nass CC, Williams AE. Trends in incidence and prevalence of major transfusion-transmissible viral infections in US blood donors, 1991 to 1996. Retrovirus Epidemiology Donor Study (REDS). JAMA. 2000 Jul 12;284(2):229-35. doi: 10.1001/jama.284.2.229. PMID 10889598
- [Background] Watanabe KK, Williams AE, Schreiber GB, Ownby HE. Infectious disease markers in young blood donors. Retrovirus Epidemiology Donor Study. Transfusion. 2000 Aug;40(8):954-60. doi: 10.1046/j.1537-2995.2000.40080954.x. PMID 10960523
- [Background] Tobler LH, Lee SR, Stramer SL, Peterson J, Kochesky R, Watanabe K, Quan S, Polito A, Busch MP. Performance of second- and third-generation RIBAs for confirmation of third-generation HCV EIA-reactive blood donations. Retrovirus Epidemiology Donor Study. Transfusion. 2000 Aug;40(8):917-23. doi: 10.1046/j.1537-2995.2000.40080917.x. PMID 10960517
- [Background] Busch MP, Watanabe KK, Smith JW, Hermansen SW, Thomson RA. False-negative testing errors in routine viral marker screening of blood donors. For the Retrovirus Epidemiology Donor Study. Transfusion. 2000 May;40(5):585-9. doi: 10.1046/j.1537-2995.2000.40050585.x. PMID 10827264
- [Background] Dinwiddie FW. Humanistic behaviorism: a model for rapprochement in residential treatment milieus. Child Psychiatry Hum Dev. 1975 Summer;5(4):254-9. doi: 10.1007/BF01433419. PMID 1139981
- [Background] Glynn SA, Smith JW, Schreiber GB, Kleinman SH, Nass CC, Bethel J, Biswas B, Thomson RA, Williams AE; Retrovirus Epidemiology Donor Study. Repeat whole-blood and plateletpheresis donors:unreported deferrable risks, reactive screening tests, andresponse to incentive programs. Transfusion. 2001 Jun;41(6):736-43. doi: 10.1046/j.1537-2995.2001.41060736.x. PMID 11399812
- [Background] Wu Y, Glynn SA, Schreiber GB, Wright DJ, Lo A, Murphy EL, Kleinman SH, Garratty G; Retrovirus Epidemiology Donor Study (REDS) Group. First-time blood donors: demographic trends. Transfusion. 2001 Mar;41(3):360-4. doi: 10.1046/j.1537-2995.2001.41030360.x. PMID 11274590
- [Background] Sanchez AM, Ameti DI, Schreiber GB, Thomson RA, Lo A, Bethel J, Williams AE; Retrovirus Epidemiology Donor Study. The potential impact of incentives on future blood donation behavior. Transfusion. 2001 Feb;41(2):172-8. doi: 10.1046/j.1537-2995.2001.41020172.x. PMID 11239218
- [Background] Liu H, Leung P, Glynn S, Murphy EL. Human T-lymphotropic virus type II RFLP subtypes a0 and b4/b5 are associated with different demographic and geographic characteristics in the United States. Virology. 2001 Jan 5;279(1):90-6. doi: 10.1006/viro.2000.0632. PMID 11145892
- [Background] Sanchez AM, Schreiber GB, Bethel J, McCurdy PR, Glynn SA, Williams AE, Gilcher R; Retrovirus Epidemiology Donor Study (REDS). Prevalence, donation practices, and risk assessment of blood donors with hemochromatosis. JAMA. 2001 Sep 26;286(12):1475-81. doi: 10.1001/jama.286.12.1475. PMID 11572740
- [Background] Glynn SA, Williams AE, Nass CC, Bethel J, Kessler D, Scott EP, Fridey J, Kleinman SH, Schreiber GB; Retrovirus Epidemiology Donor Study. Attitudes toward blood donation incentives in the United States: implications for donor recruitment. Transfusion. 2003 Jan;43(1):7-16. doi: 10.1046/j.1537-2995.2003.00252.x. PMID 12519425
- [Background] Schreiber GB, Glynn SA, Damesyn MA, Wright DJ, Tu Y, Dodd RY, Murphy EL; Retrovirus Epidemiology Donor Study. Lapsed donors: an untapped resource. Transfusion. 2003 Jan;43(1):17-24. doi: 10.1046/j.1537-2995.2003.00290.x. PMID 12519426
- [Background] Sanchez AM, Schreiber GB, Glynn SA, Bethel J, Kessler D, Chang D, Zuck TF; Retrovirus Epidemiology Donor Study. Blood-donor perceptions of health history screening with a computer-assisted self-administered interview. Transfusion. 2003 Feb;43(2):165-72. doi: 10.1046/j.1537-2995.2003.00295.x. PMID 12559011
- [Background] Sharma UK, Stramer SL, Wright DJ, Glynn SA, Hermansen S, Schreiber GB, Kleinman SH, Busch MP; Retrovirus Epidemiology Donor Study. Impact of changes in viral marker screening assays. Transfusion. 2003 Feb;43(2):202-14. doi: 10.1046/j.1537-2995.2003.00291.x. PMID 12559016
- [Background] Busch MP, Kleinman SH, Nemo GJ. Current and emerging infectious risks of blood transfusions. JAMA. 2003 Feb 26;289(8):959-62. doi: 10.1001/jama.289.8.959. No abstract available. PMID 12597733
- [Background] Wang B, Schreiber GB, Glynn SA, Nass CC, Smith JW, Higgins MJ, Hutching ST, Wright DJ, McEntire RL, Murphy EL; Retrovirus Epidemiology Donor Study. Prevalence of transfusion-transmissible viral infections in first-time US blood donors by donation site. Transfusion. 2003 Jun;43(6):705-12. doi: 10.1046/j.1537-2995.2003.00399.x. PMID 12757520
- [Background] Glynn SA, Busch MP, Schreiber GB, Murphy EL, Wright DJ, Tu Y, Kleinman SH; NHLBI REDS Study Group. Effect of a national disaster on blood supply and safety: the September 11 experience. JAMA. 2003 May 7;289(17):2246-53. doi: 10.1001/jama.289.17.2246. PMID 12734136
- [Background] Schreiber GB, Sanchez AM, Glynn SA, Wright DJ; Retrovirus Epidemiology Donor Study. Increasing blood availability by changing donation patterns. Transfusion. 2003 May;43(5):591-7. doi: 10.1046/j.1537-2995.2003.00388.x. PMID 12702179
- [Background] Roback JD, Drew WL, Laycock ME, Todd D, Hillyer CD, Busch MP. CMV DNA is rarely detected in healthy blood donors using validated PCR assays. Transfusion. 2003 Mar;43(3):314-21. doi: 10.1046/j.1537-2995.2003.00312.x. PMID 12675715
- [Background] Sacher RA, Luban NL, Ameti DI, Friend S, Schreiber GB, Murphy EL. Low prevalence of flower cells in U.S.A. blood donors infected with human T-lymphotrophic virus types I and II. Br J Haematol. 1999 Jun;105(3):758-63. doi: 10.1046/j.1365-2141.1999.01408.x. PMID 10354142
- [Background] Guiltinan AM, Murphy EL, Horton JA, Nass CC, McEntire RL, Watanabe K. Psychological distress in blood donors notified of HTLV-I/II infection. Retrovirus Epidemiology Donor Study. Transfusion. 1998 Nov-Dec;38(11-12):1056-62. doi: 10.1046/j.1537-2995.1998.38111299056317.x. PMID 9838938
- [Background] Kleinman S, Busch MP, Hall L, Thomson R, Glynn S, Gallahan D, Ownby HE, Williams AE. False-positive HIV-1 test results in a low-risk screening setting of voluntary blood donation. Retrovirus Epidemiology Donor Study. JAMA. 1998 Sep 23-30;280(12):1080-5. doi: 10.1001/jama.280.12.1080. PMID 9757856
- [Background] Murphy EL, Glynn S, Watanabe K, Fridey J, Smith J, Sacher R, Wright D, Schreiber G, Luban N. Laboratory test differences associated with HTLV-I and HTLV-II infection. Retrovirus Epidemiology Donor Study Investigators. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Apr 1;17(4):332-8. doi: 10.1097/00042560-199804010-00007. PMID 9525434
- [Background] Thomson RA, Bethel J, Lo AY, Ownby HE, Nass CC, Williams AE. Retention of "safe" blood donors. The Retrovirus Epidemiology Donor Study. Transfusion. 1998 Apr;38(4):359-67. doi: 10.1046/j.1537-2995.1998.38498257374.x. PMID 9595018
- [Background] Damesyn MA, Glynn SA, Schreiber GB, Ownby HE, Bethel J, Fridey J, McMullen Q, Garratty G, Busch MP; NHLBI Retrovirus Epidemiology Donor Study. Behavioral and infectious disease risks in young blood donors: implications for recruitment. Transfusion. 2003 Nov;43(11):1596-603. doi: 10.1046/j.1537-2995.2003.00532.x. PMID 14617320
- [Background] Pellett PE, Wright DJ, Engels EA, Ablashi DV, Dollard SC, Forghani B, Glynn SA, Goedert JJ, Jenkins FJ, Lee TH, Neipel F, Todd DS, Whitby D, Nemo GJ, Busch MP; Retrovirus Epidemiology Donor Study. Multicenter comparison of serologic assays and estimation of human herpesvirus 8 seroprevalence among US blood donors. Transfusion. 2003 Sep;43(9):1260-8. doi: 10.1046/j.1537-2995.2003.00490.x. PMID 12919429
- [Background] Rugege-Hakiza SE, Glynn SA, Hutching ST, Bethel J, Nass CC, McEntire RL, Hirschler NV, Campbell JG, Ladavac A, Schreiber GB; Retrovirus Epidemiology Donor Study. Do blood donors read and understand screening educational materials? Transfusion. 2003 Aug;43(8):1075-83. doi: 10.1046/j.1537-2995.2003.00473.x. PMID 12869113
- [Background] Kleinman SH, Kuhns MC, Todd DS, Glynn SA, McNamara A, DiMarco A, Busch MP; Retrovirus Epidemiology Donor Study. Frequency of HBV DNA detection in US blood donors testing positive for the presence of anti-HBc: implications for transfusion transmission and donor screening. Transfusion. 2003 Jun;43(6):696-704. doi: 10.1046/j.1537-2995.2003.00391.x. PMID 12757519
- [Background] Schreiber GB, Sanchez AM, Garratty G, Nass CC, Tu Y, Busch MP; Retrovirus Epidemiology Donor Study. Mammalian brain consumption by blood donors in the United States: brains today, deferred tomorrow? Transfusion. 2004 May;44(5):667-74. doi: 10.1111/j.1537-2995.2004.03114.x. PMID 15104646
- [Background] Busch MP, Glynn SA, Stramer SL, Strong DM, Caglioti S, Wright DJ, Pappalardo B, Kleinman SH; NHLBI-REDS NAT Study Group. A new strategy for estimating risks of transfusion-transmitted viral infections based on rates of detection of recently infected donors. Transfusion. 2005 Feb;45(2):254-64. doi: 10.1111/j.1537-2995.2004.04215.x. PMID 15660836
- [Background] Tobler LH, Bianco C, Glynn SA, Schreiber GB, Dille BJ, Prince HE, Lanciotti RS, Linnen JM, Gallarda J, Shyamala V, Smith D, Kleinman SH, Busch MP; NHLBI Retrovirus Epidemiology Study (REDS). Detection of West Nile virus RNA and antibody in frozen plasma components from a voluntary market withdrawal during the 2002 peak epidemic. Transfusion. 2005 Apr;45(4):480-6. doi: 10.1111/j.0041-1132.2005.04266.x. PMID 15819666
- [Background] Kleinman S, Glynn SA, Busch M, Todd D, Powell L, Pietrelli L, Nemo G, Schreiber G, Bianco C, Katz L; NHLBI Retrovirus Epidemiology Study (REDS). The 2003 West Nile virus United States epidemic: the America's Blood Centers experience. Transfusion. 2005 Apr;45(4):469-79. doi: 10.1111/j.0041-1132.2005.04315.x. PMID 15819665
- [Background] Kleinman SH, Glynn SA, Higgins MJ, Triulzi DJ, Smith JW, Nass CC, Garratty G, Murphy EL, LeParc GF, Schreiber GB, King MR, Chamberland ME, Nemo GJ. The RADAR repository: a resource for studies of infectious agents and their transmissibility by transfusion. Transfusion. 2005 Jul;45(7):1073-83. doi: 10.1111/j.1537-2995.2005.00171.x. PMID 15987350
- Available data/document: Operations Manual: REDS-GSR/GLPR — http://biolincc.nhlbi.nih.gov/studies/gsrglpr/ — Samples and characterization data. NHLBI provides controlled access to samples through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a materials use agreement.
- Available data/document: Individual Participant Data Set: REDS-HTLV — http://biolincc.nhlbi.nih.gov/studies/reds/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms: REDS-HTLV — http://biolincc.nhlbi.nih.gov/studies/reds/
- Available data/document: Operations Manual: REDS-RADAR — http://biolincc.nhlbi.nih.gov/studies/radar/ — Samples and characterization data. NHLBI provides controlled access to samples through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a materials use agreement.